CLINICAL TRIAL: NCT05434637
Title: Developing Tools and a Care Path for Somatosensory Tinnitus
Brief Title: Somatosensory Tinnitus RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C3924-R
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Tinnitus
Keywords: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Physical Therapy Modalities; Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Individualized Physiotherapy (Experimental): Individuals randomized to this group will receive physical therapy, personalized for the participant's specific needs, and include exercises to be performed at home.
  Interventions: Other: Physical Therapy
- Sound-based Therapy (Active Comparator): Individuals randomized to this group will receive sound-based therapy, consistent with an audiology-based standard of care treatment.
  Interventions: Other: Sound-based Therapy
- Combination Therapy (Experimental): Individuals randomized to this group will receive both individualized physical therapy and sound-based therapy.
  Interventions: Other: Combination Therapy

INTERVENTIONS:
Other: Physical Therapy — Individuals randomized to this intervention will receive physical therapy, personalized for the participant's specific needs, and include exercises to be performed at home.
  Other Names: Individualized Physiotherapy
  Arms: Individualized Physiotherapy
Other: Sound-based Therapy — Individuals randomized to this intervention will receive sound-based therapy, consistent with an audiology-based standard of care treatment.
  Other Names: Audiology Therapy
  Arms: Sound-based Therapy
Other: Combination Therapy — Individuals randomized to this intervention will receive both individualized physical therapy and sound-based therapy.
  Other Names: Physical Therapy + Audiology Therapy
  Arms: Combination Therapy

SUMMARY:
The purpose of this study is to learn more about a type of tinnitus (ringing in the ears) known as "somatosensory tinnitus." This type of tinnitus is suspected when the tinnitus perception changes following head and/or neck movements. This study is also exploring a possible way to treat somatosensory tinnitus.

DETAILED DESCRIPTION:
The purpose of this study is to: (1) develop a screening tool for somatosensory tinnitus and (2) perform a randomized clinical trial comparing different treatment approaches for somatosensory tinnitus. The investigators want to find out if individualized physical therapy, alone or in combination with audiology-based sound therapy, is beneficial for treating somatosensory tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* Constant, chronic tinnitus (6-months in duration)
* bothersome tinnitus based on TFI score and self-reported loudness
* able to modulate tinnitus perception with head, neck, and/or jaw maneuvers

Exclusion Criteria:

* Middle ear pathology
* not a candidate for physical therapy
* injury to the temporomandibular area in past 3 months
* active pathology in the orofacial region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in TFI Score | Measured at at baseline; 8 and 12 weeks post-randomization
  The TFI is a 25-item questionnaire that evaluates treatment responsiveness (i.e., changes in functional effects of tinnitus over time). Total possible score ranges from 0-to-100 (scores >25 indicate tinnitus is a significant problem).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Theodoroff, PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No